CLINICAL TRIAL: NCT00709930
Title: Randomized Placebo-Controlled Trial of Efficacy and Safety of Weak Extremely Low Frequency Electromagnetic Field in Mild and Moderate Essential Hypertension
Brief Title: Efficacy and Safety of Weak Extremely Low Frequency Electromagnetic Fields in Mild and Moderate Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyoto University (Other)
Responsible Party: Masanori Fukushima, Translarional Research center
Organization: Kyoto University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MF-II-01
Record Dates: First submitted 2008-06-27; First posted 2008-07-03 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1,Exposed to ELF-EMF (Active Comparator): Device: Magnetic field generator Exposure to 1-μT 8/6-Hz ELF-EMF
  Interventions: Device: Magnetic field generator
- 2,Placebo (Placebo Comparator): Device: Placebo device with no magnetic fields
  Interventions: Device: Placebo magnetic field generator

INTERVENTIONS:
Device: Magnetic field generator — dosage:Magnetic field generator Exposure to 1-μT 8/6-Hz ELF-EMF frequency:10min/day duration:1 month
  Arms: 1,Exposed to ELF-EMF
Device: Placebo magnetic field generator — Placebo device with no magnetic fields
  Arms: 2,Placebo

SUMMARY:
This study will evaluate the efficacy and safety of weak extremely low frequency electromagnetic fields (ELF-EMF) in mild and moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 20 years to 74 years
* Genders : Both
* The severity of hypertension: mild and moderate (WHO/ISH criteria stage I-II) Systolic blood pressure (SBP) >/= 140 and/or diastolic blood pressure (DBP)>/= 90 (untreated hypertension cases)

Exclusion Criteria:

* Any of the following medical conditions:
* Severe essential hypertension (DBP >110)
* Secondary or malignant hypertension
* History or symptoms of cerebral vascular disease
* History of myocardial infarction
* History of angina pectoris, atrial fibrillation, heart failure and arrhythmia
* Renal dysfunction (serum creatinine > 2.1mg/dl)
* Severe hepatic dysfunction
* Uncontrolled diabetes
* Allergy, drug sensitivity or chronic skin disease
* Peptic ulcer disease
* Current pregnancy or lactation
* Depression that needs to be treated
* Hypertension controlled with antihypertensive medication

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The difference between the ELF-EMF and sham groups with respect to the absolute change in SBP value between baseline and the end of the exposure regimen (the age of the pre-exposure values for the last two sessions). | baseline and the end of the exposure regimen (the average of the pre-exposure values for the last two sessions)

SECONDARY OUTCOMES:
The difference between the ELF-EMF and sham groups with respect to the change in DBP value between baseline and the end of the exposure regimen (the average of the pre-exposure values for the last two sessions) | baseline and the end of the exposure regimen (the average of the pre-exposure values for the last two sessions)
The change in both SBP and DBP values between pre-exposure and post-exposure for each session (averaged over the regimen) | for each session
The incidence of adverse events | during exposure and at the end of the exposure period and at six months after exposure

CONTACTS AND LOCATIONS:
Overall Officials: Masanori Fukushima, Principal Investigator — Kyoto University Hospital
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan